CLINICAL TRIAL: NCT03574909
Title: Investigating the Role of Early Low-dose Aspirin in Diabetes: A Phase III Multicentre Double-blinded Placebo-controlled Randomised Trial of Low-dose Aspirin Initiated in the First Trimester of Diabetes Pregnancy
Brief Title: IRELAnD: Investigating the Role of Early Low-dose Aspirin in Diabetes
Acronym: IRELAnD
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Royal College of Surgeons, Ireland (Other)
Collaborators: Health Research Board, Ireland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Ireland-Rct-v1-0218; 2018-000770-29 (EudraCT Number)
Record Dates: First submitted 2018-03-15; First posted 2018-07-02 (Actual); Last update posted 2018-08-27 (Actual); Status verified 2018-03

CONDITIONS: Pre-Gestational Diabetes
MeSH Terms: interventions — Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment Arm (Experimental): Treatment Arms: Tromalyt® 150mg prolong release capsule for oral ingestion. The capsule contains 150mg of anti-platelet agent acetylsalicylic acid, maize starch and Sucrose 20:80. The capsule also contains Copovidone (Kollidon VA-64), Eudragit L, Ethylcellulose and Triacetin. The capsule is made with gelatin, erythrosine, quinoline yellow, titanium dioxide. Tromalyt® is trademark of Meda Pharma SL (Reg 59.210).
  There is no requirement for the first dose to be administered in the clinic under observation.
  The dosing frequency is once daily. Subjects will be instructed to take the study medication at the same time each day.
  No specific precautions are required in relation to concomitant food intake.
  Interventions: Drug: Aspirin
- Control Arm (Placebo Comparator): Placebos to be used are hard gelatin capsules (Sanitatis®) for patients randomized to the placebo arm. These capsules are externally identical to Tromalyt capsule. The capsules contain 198mg microcrystalline cellulose and 2mg of magnesium stearate (Sanitatis®) Placebo: There is no requirement for the first dose to be administered in the clinic under observation.
  The dosing frequency is once daily. Subjects will be instructed to take the study medication at the same time each day.
  No specific precautions are required in relation to concomitant food intake.
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Aspirin — Tromalyt® 150mg prolong release capsule for oral ingestion. The capsule contains 150mg of anti-platelet agent acetylsalicylic acid, maize starch and Sucrose 20:80. The capsule also contains Copovidone (Kollidon VA-64), Eudragit L, Ethylcellulose and Triacetin. The capsule is made with gelatin, erythrosine, quinoline yellow, titanium dioxide.
  Other Names: Tromalyt
  Arms: Treatment Arm
Drug: Placebos — Size 0 hard gelatin capsules containing 99% of microcrystalline cellulose and 1% of magnesium stearate (Sanitatis®). The capsules contain 198mg microcrystalline cellulose and 2mg of magnesium stearate
  Other Names: Sanitatis
  Arms: Control Arm

SUMMARY:
To investigate the effect of aspirin therapy initiated in the first trimester of pregnancy in women with pregestational type I or type II diabetes on a composite clinical measure of placental dysfunction (preeclampsia, preterm birth less than 34 weeks, birthweight below the 10th centile or perinatal mortality).

DETAILED DESCRIPTION:
Pregestational diabetes represents a high-risk for evolution of preeclampsia (PET), with rates of PET within this group at approximately 20%. The combination of diabetes and preeclampsia places the pregnancy at heightened risk for hypoxia and stillbirth. Placental dysfunction, due to disordered early placental development, is central to the disease process. Early placental disease is followed months later by clinical manifestations of PET, which reflect widespread endothelial dysfunction resulting in vasoconstriction, ischaemia and increased vascular permeability. While not all adverse perinatal outcomes in diabetes are attributed to placental dysfunction, any therapy that offers the potential to optimise placentation in this group deserves close attention.

The dose of aspirin used in randomized trials ranges from 50mg to 150mg. For some women, particularly those with type 2 diabetes-related obesity, the commonly-used 60mg dose may be too low to exert a full effect on thromboxane production. Recent work by one of the collaborators for this submission indicates that 20% of patients in Ireland with established coronary artery disease are inadequately 'protected' by aspirin, as evidenced by a thromboxane B2 level of >2.2 (indicating platelet aggregation of greater than 20%). Age, hypertension and weight were identified as risk factors for an inadequate aspirin response. Furthermore, randomized trials of this nature are potentially compromised by an inability to confidently ensure patient compliance. The use of platelet function assays for a sub-group of the participants in this proposed work offers the potential both to determine whether body mass index and gestational age influence the ability to achieve an optimal biologic drug effect and also to confirm patient compliance.

Pre-pregnancy nephropathy places a woman at particularly high risk for superimposed preeclampsia and for fetal growth restriction. Microalbuminuria is known to be the forerunner for diabetic nephropathy. Indeed, microalbuminuria is considered to be a marker of generalized endothelial dysfunction. Whether sub-threshold degrees of microvascular disease, as evidenced by microalbuminuria in early gestation, may confer a heightened risk of preeclampsia, is unclear. Furthermore, whether aspirin therapy may benefit this subgroup with microalbuminuria has not been studied. The largest study to date to investigate the prevalence of microalbuminuria was conducted in Denmark, on a cohort of 1,200 pregnant women with type I diabetes and documented a fourfold increase in risk of developing preeclampsia among microalbuminuric women compared to normoalbuminuric diabetic women. A secondary analysis of the MFMU aspirin study documented no increased risk of preeclampsia among women with diabetes who had proteinuria <499mg/24h in early pregnancy. A randomized trial of aspirin therapy for the prevention of placental dysfunction in the setting of pregestational diabetes may clarify whether aspirin therapy confers particular benefit among microalbuminuric women.

Importantly, although NICE has issued guidance on the prevention of hypertension in pregnancy that includes a recommendation that women deemed to be at high risk for hypertension in pregnancy be considered for low-dose aspirin after 12 weeks' gestational age, and pregestational diabetes is listed as an example of 'high risk', this recommendation is not supported by randomized-trial evidence demonstrating a benefit to aspirin therapy in women with diabetes. Furthermore, this guidance is at variance with international guidelines on the management of diabetes in pregnancy, none of which includes a recommendation that aspirin is prescribed to this group. This reflects the dearth of studies that have been done on this high-risk subgroup and the paucity of evidence gleaned from meta analyses in favour of aspirin therapy in this group.

Routine prescription of aspirin therapy for women with pre-existing diabetes does not represent standard care in Ireland. The Mother and Baby CTN is well placed to answer the clinical question here, centred on whether low-dose antiplatelet therapy in pregnancy may carry the potential to optimise pregnancy outcome in this high-risk group.

9.2 Preclinical data Aspirin is a non-steroidal anti-inflammatory drug (NSAID) with analgesic and antipyretic effects. Aspirin also inhibits cyclo-oxygenase isoforms 1 and 2 (COX1/COX2) by irreversible acetylation, thus inhibiting the biosynthesis of prostaglandins and thromboxanes from arachadonic acid. Aspirin's antiplatelet effects relate to its inhibition of the production of platelet thromboxane A2, a prothrombotic vasoconstrictor. This inhibitory effect is cumulative on repeat dosing, with complete suppression of platelet thromboxane synthesis estimated to occur within a few days after daily dosing of 20 to 50mg and more rapid suppression occurring with larger doses of 150-300mg. Much higher doses are required for anti-inflammatory, analgesic and antipyretic effects (3.6-4g daily).

Animal studies showed that at very large dose levels, aspirin is teratogenic in rodents, with cranial defects, neural tube defects, and cardiac defects among the most consistent findings. Offspring of food-restricted rats that also received aspirin 250 mg/kg/day had more than twice the incidence of malformations as those that received aspirin without food restriction. The most notable malformations were rib and limb defects and umbilical hernias. At higher dose levels, aspirin produced similar embryotoxicity in rhesus monkeys. The anomalies observed included neural tube defects, skeletal malformations, and facial clefts. A 2003 review of the experimental animal literature noted diaphragmatic hernia, ventricular septal defect, or midline defects associated with aspirin or other NSAIDs. This analysis noted that the general quality of available reports was poor, but work in rats, with bolus administration of the maximum tolerable dose of aspirin, as well as some reversible COX-1 inhibitors, consistently produced midline and cardiac defects. In rabbits, because of maternal toxicity, aspirin cannot be administered at high enough dose levels to produce developmental defects.

9.3 Clinical data Low-dose aspirin has been investigated for the prevention of preeclampsia owing to its negative effect on thromboxane production. An imbalance between prostacyclin and thromboxane plays a key role in the development of PET and is believed to result from shallow placental invasion and ischaemia that occur shortly after implantation, very early in the first trimester of pregnancy.

Studies on the role of aspirin in the prevention of preeclampsia in high-risk women have yielded conflicting results. Initial studies suggested a protective effect. Subsequently, some larger studies failed to identify a benefit to aspirin therapy although CLASP did demonstrate a benefit in women affected by early-onset severe preeclampsia in a prior pregnancy.

A metaanalysis, based on 27 trials on 31,678 women, concluded that aspirin is effective in preventing preeclampsia, although the effect, a 10% reduction in PET incidence, was too modest to warrant routine use in all women. The authors concluded that 'Despite a very large dataset, the evidence base for particular groups of high risk women remains limited '. Pre-existing diabetes was identified in 905 randomized women in this metaanalysis and the authors calculated a relative risk for PET of 0.76 (CI 0.56 to 1.04), thus failing to demonstrate a statistically significant effect. No information is provided on gestational age at recruitment for this subanalysis, but very few studies were included that recruited women <16 weeks. Two thirds of the overall dataset were recruited after 20 weeks' gestational age. However, if started early in pregnancy the treatment may be effective, although studies are few and results are inconsistent, demonstrated a 17% reduction in the incidence of PET when combining studies of different design. These authors stratified patients according to risk-status for PET and concluded that aspirin may confer a 25% reduction in preeclampsia for women deemed to be at high risk for developing the disease. Pre-pregnancy diabetes constituted a high risk factor in this analysis. However, any benefit of aspirin therapy in reducing the incidence of PET in this group was not demonstrated by the Askie metaanalysis.

Few studies investigate the role of aspirin in preventing preeclampsia specifically in women with diabetes. Only two randomized trials have recruited women with pregestational diabetes without chronic hypertension or established renal disease. A large multicenter MFMU Network study investigated the role of aspirin in prevention of PET for high-risk women, which included a subgroup of 471 women with pregestational diabetes. Although this study did not demonstrate a difference in the incidence of PET between aspirin and placebo groups, women were recruited in the 2nd trimester (mean GA at recruitment 18 weeks +/- 4 weeks). It is plausible that any effect of aspirin on placentation may only be observed if therapy is initiated in the first trimester. Indeed, a recent metaanalysis investigating the role of aspirin in prevention of perinatal death concludes that low-dose aspirin has potential to reduce perinatal mortality when initiated prior to 16 weeks compared to later treatment. Therefore, if aspirin is to be used for the prevention of placental dysfunction, it must be initiated before the second active phase of trophoblast invasion, which takes place from 14 weeks' gestation onwards. No randomized trials investigating the role of aspirin in prevention of preeclampsia have initiated treatment in the first trimester, the gestational period at which it is most likely to exert an effect on placentation.

9.4 Rationale and risks/benefits The investigational medicinal product to be used in this trial: Tromalyt® 150mg prolong release capsule for oral ingestion. The gelatine capsule contains 150mg of anti-platelet agent acetylsalicylic acid, maize starch and Sucrose 20:80. . Tromalyt® is trademark of Meda Pharma SL (Reg 59.210).

Placebo hard gelatin capsules (Sanitatis®) will be used for patients randomized to the placebo arm. These capsules are externally identical to Tromalyt capsule. The capsules contain 198mg microcrystalline cellulose and 2mg of magnesium stearate (Sanitatis®)

. The antiplatelet properties of aspirin may confer a beneficial effect on placental function, owing to the putative imbalance between thromboxane and prostacyclin that are thought to result in shallow placental invasion in the first trimester. The ability of antiplatelet therapy such as aspirin to potentially optimize placental architecture early in pregnancy may lead to a greater prospect of a low-resistance placental circulation being established early in pregnancy in this cohort of women with microangiopathic disease relating to pre-pregnancy diabetes. Therefore, the study hypothesis is that initiation of low-dose aspirin in the first trimester of pregnancy may lead to a reduction in placental dysfunction-mediated adverse perinatal outcome (namely, pre-eclampsia, fetal growth restriction, preterm birth or perinatal death).

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy with a pre-pregnancy diagnosis of type I or type II diabetes of at least 6 months' duration

Exclusion Criteria:

* • Aspirin hypersensitivity (prior bronchospasm/ urticarial/ angioedema with aspirin)

  * Peptic ulcer disease
  * Known bleeding diathesis
  * Multifetal gestation
  * Severe early-onset preeclampsia in a previous pregnancy
  * Patient already on aspirin
  * Established chronic renal disease/ macroalbuminuria
  * Chronic hypertension (antihypertensive therapy in first trimester)
  * Current selective serotonin reuptake inhibitor (SSRI) use (or SSRI use within 7 days)
  * Inability to speak or read English
  * Age less than 18 years
  * Use of any other investigational medicinal product within previous 30 days
  * Presence of any illness or condition that might interfere with the patient's ability to comply with the study procedures

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2018-09 (Estimated); Primary Completion 2021-09 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Preeclampsia - Change in blood pressure (Hypertension) | From 20 weeks gestation to delivery
  (i) greater than or equal to 140mmHg systolic or greater than or equal to 90mmHg diastolic on two occasions at least 4 hours apart after 20 weeks' gestation in a woman with a previously normal blood pressure.
  Or (ii) greater than or equal to 160mmHg systolic or greater than or equal to 110mmHg diastolic (such hypertension can be confirmed within a short interval (minutes) to facilitate timely antihypertensive therapy.perinatal mortality
Preeclampsia - Change in Proteinuria | From 20 weeks gestation to birth
  Greater than or equal to 300mg per 24-hour urine collection, or a urinary protein: creatinine ratio greater than or equal to 0.3 or +3 proteinuria on dipstick urinalysis.
Birth weight | weight will be measured on the day of birth and plotted on standard WHO UK RCPCH growth charts (per gender).
  Birth weight less than the 10th percentile for gestational age:
Preterm birth | Gestational age at birth will be verified with respect to the Estimated Date of Delivery calculated at the first study visit.
  -Preterm birth less than 34+0 weeks:
Perinatal mortality | Stillbirth or neonatal death after 24 completed weeks of gestation and within 28 days of birth.
  Perinatal mortality

SECONDARY OUTCOMES:
Parameters of neonatal morbidity: Gestational age at delivery | recorded at the time of birth, in weeks and days post Last Menstrual Period, or in accordance with ultrasound-derived gestational age, as above
  Gestational age at delivery
Parameters of neonatal morbidity: Birth weight | recorded (in grams) on the day of birth)
  Birth weight
Parameters of neonatal morbidity: NICU admission | Up to 10 days post birth
  NICU admission
Respiratory morbidity: Duration of invasive ventilation | Up to 6 weeks after birth
  Duration of invasive ventilation
Duration of O2 | Up to 6 weeks after birth
  Respiratory morbidity: Duration of O2
Duration of hospital stay | Up to 6 weeks after birth
  Respiratory morbidity: Duration of hospital stay
Use of nitric oxide | Up to 6 weeks after birth
  Respiratory morbidity: Use of nitric oxide
Number and type of inotropes | Up to 6 weeks after birth
  Respiratory morbidity: Number and type of inotropes
Duration of inotrope use | Up to 6 weeks after birth
  Respiratory morbidity: Duration of inotrope use
Apgar score | Apgar score will be recorded within 5 minutes of birth, as per standard clinical care.
  Apgar score <7 at 5 minutes
Umbilical artery acidosis at birth | measured where clinically indicated at birth
  Umbilical arterial pH and acid-base status will be measured where clinically indicated at birth (namely in an infant born in the setting of suspected perinatal compromise). In addition to cord pH, the first infant pH will also be recorded, if obtained.
Intracranial haemorrhage: | measured where clinically indicated at birth
  Evidence of bleeding within the intraventricular or periventricular areas of the neonatal brain, identified with cranial ultrasound or alternate imaging.
Culture-proven sepsis: | measured where clinically indicated at birth
  A diagnosis of neonatal sepsis will be made when appropriate clinical features are confirmed by positive microbiological cultures.
Necrotising enterocolitis | measured where clinically indicated at birth
  Defined as presence of radiologic signs (Bell Stage II or greater).
Hypoxic ischaemic encephalopathy | measured where clinically indicated at birth
  A diagnosis of hypoxic ischemic encephalopathy will be recorded where the following criteria are met:
  * Apgar score ≤5 at 10 minutes after birth
  * Continued need for endotracheal or mask ventilation at 10 minutes after birth
  * Acidosis within 60 minutes of birth (defined as any occurrence of umbilical cord arterial or capillary pH <7.0 or a base deficit ≥16mmol/L)
  * And/ or clinical seizures or moderate to severe encephalopathy using the Sarnat grading system
Shoulder dystocia | birth
  Shoulder dystocia is defined as a vaginal cephalic delivery that requires additional obstetric manoeuvres to deliver the fetus after the head has delivered and gentle traction has failed
Composite measure of Maternal outcomes not directly related to primary outcome | Delivery
  Mode of delivery: Recorded on day of delivery, as follows:
  Spontaneous vaginal birth (with spontaneous onset of labour) Spontaneous vaginal birth (with induction of labour) Assisted vaginal birth (forceps) with spontaneous onset of labour Assisted vaginal birth (forceps) with induction of labour Assisted vaginal birth (ventouse) with spontaneous onset of labour Assisted vaginal birth (ventouse) with induction of labour Emergency intrapartum Caesarean section with induction of labour Emergency intrapartum Caesarean section with spontaneous onset of labour Emergency pre-labour Caesarean section (i.e. unscheduled) Elective Caesarean section (scheduled) Elective Caesarean section with spontaneous onset of labour
Haemorrhage: | During birth
  Loss of 500ml of blood or more from the genital tract within 24 hours of delivery. Peripartum blood loss will be recorded as average or excessive (500ml or more) for all deliveries. In addition, requirement for the following measures to reduce peripartum blood loss will be recorded:
  Oxytocin 10IU, oxytocin infusion, ergometrine, syntometrine, hemabate, misoprostol, intrauterine balloon tamponade, B-Lynch suture, interventional radiologic manoeuvres, hysterectomy, blood transfusion (including number and nature of blood products)
Sepsis | During birth
  Culture-proven infection in addition to systemic manifestations of infection

REFERENCES:
- [Derived] Finnegan C, Dicker P, Asandei D, Higgins M, O'Gorman N, O' Riordan M, Dunne F, Gaffney G, Newman C, McAuliffe F, Ciprike V, Fernandez E, Malone FD, Breathnach FM. The IRELAnD study-investigating the role of early low-dose aspirin in diabetes mellitus: a double-blinded, placebo-controlled, randomized trial. Am J Obstet Gynecol MFM. 2024 Apr;6(4):101297. doi: 10.1016/j.ajogmf.2024.101297. Epub 2024 Mar 8. PMID 38461094